CLINICAL TRIAL: NCT04558710
Title: The Effect of Frequent Continuous Glucose Monitoring Use on Glucose Variability in Preschoolers With Type 1 Diabetes - The VibRate Study
Brief Title: The Effect of Frequent Continuous Glucose Monitoring Use on Glucose Variability in Preschoolers With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: International Society for Pediatric and Adolescent Diabetes (Unknown); Kinderkrankenhaus auf der Bult, Hannover, Germany (Unknown); Department of Pediatrcs, Endocrinology and Diabetes Medical University of Silesia in Katowice, Poland (Unknown); Pediatric Diabetes and Metabolic Disorders Unit, Regional Center for Pediatric Diabetes, University City Hospital of Verona, Verona, Italy (Unknown); Yale University School of Medicine, Department of Pediatrics, New Haven, Connecticut, United States (Unknown); Pediatric Endocrinology Unit, Paediatrics Department, Maternal and Paediatrics Centre, São João University and Hospital Centre, Porto, Porto, Portugal (Unknown); Department of Pediatrics, Section on Diabetes and Metabolism, V. Buzzi Children's Hospital, University of Milan, Milan, Italy (Unknown); Pediatric Endocrinology Unit. Hospital Pediátrico. Centro Hospitalar e Universitário de Coimbra. Coimbra. Portugal (Unknown); Diaboss, Amsterdam, Netherlands (Unknown); Medical School, University of Valparaiso, San Felipe, Chile. (Unknown); Department of Pediatric Endocrinology and Diabetes, Koç University Hospital, İstanbul, Turkey. (Unknown); University of Roma La Sapienza (Other); Department of Pediatrics, San Raffaele Scientific Institute , Milan, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: VibRate Study
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2020-09

CONDITIONS: Type 1 Diabetes; Continuous Glucose Monitoring; Children; Glucose Variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CGM: CGM users
- SMBG: Non-CGM users

SUMMARY:
The purpose of this study is to determine whether continuous glucose monitoring will improve glucose variability as measured by the coefficient of variation of glucose levels in very young children with T1D. The study adopts an open-label, multi-centre, multinational, prospective registry-based population cohort design contrasting CGM use to SMBG alone in young children with type 1 diabetes over 12 months.

The primary endpoint is the difference between treatment modalities (CGM vs SMBG alone) in glycaemic variability, measured as the coefficient of variation of glucose levels, during the 12 months observational period. Other Key edpoints include time in range 70-180 mg/dl, time below range 70 mg/dl and time above range 180 mg/dl.

ELIGIBILITY:
Key inclusion criteria:

1. Age below 7 years of age (at inclusion)
2. Type 1 diabetes for at least 6 months
3. Insulin pump user for at least 3 months
4. Treated with rapid or ultra-rapid acting insulin analogue

Key exclusion criteria:

1. Physical or psychological disease likely to interfere with normal conduct of the study
2. Untreated coeliac disease or thyroid disease
3. Current treatment with drugs known to interfere with glucose metabolism
4. Subject/carer's severe visual impairment
5. Subject/carer's severe hearing impairment

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pre-school children below age of 7 years with type 1 diabetes (for at least 6 months) and treated with insulin pump fo at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation | 1 year

SECONDARY OUTCOMES:
Time in Range | 1 year
  Time in Range 70 - 180 mg/dl
Time Above Range | 1 year
  Time in Range above 180 mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty - University of Ljubljana, Ljubljana, Slovenia